CLINICAL TRIAL: NCT06860711
Title: Safety of Short-term NSAID Use in the Postoperative Setting in Pediatric Patients With Chronic Kidney Disease
Brief Title: Safety of Short-course of NSAIDs in Pediatric Patients With CKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-1252
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease; Pediatric Urology
Keywords: NSAIDs; CKD; Pediatrics; Urology; post-surgical
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NSAID (Experimental): Participants will receive an intravenous (IV) ketorolac 0.5mg/kg/dose, 15mg maximum, for no more than 8 doses in keeping with the investigators' routine clinical practice. Participants will then receive the oral (PO) ibuprofen suspension 10mg/kg/dose, 400mg maximum. The total duration of intervention (IV + PO) will not exceed 5 days.
  Interventions: Drug: NSAIDs
- Placebo (Placebo Comparator): The IV formulation will be Normal Saline. The PO formulation will be compounded to have a similar look, volume, consistency and taste to the experimental medication. Participants will receive the IV formulation for no more than 8 doses. Participants will then receive the PO formulation. The total duration of intervention (IV + PO) will not exceed 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NSAIDs — IV formulation: ketorolac 0.5mg/kg/dose, 15mg maximum, no more than 8 doses total PO formulation: ibuprofen suspension 10mg/kg/dose, 400mg maximum Total duration (IV + PO) will not exceed 5 days.
  Arms: NSAID
Drug: Placebo — IV or PO medication, compounded to have similar look, consistency and taste to the corresponding medications
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if non-steroidal anti-inflammatory (NSAID) use in the postoperative setting increases the risk of acute kidney injury (AKI) in pediatric patients with mild-to-moderate chronic kidney disease (CKD). The investigators hypothesize that there is no increased risk. This will be a limited pilot study within a Pediatric Urology population, intended to inform future work in a larger patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 months of age
* diagnosis of CKD stages 2-3a, confirmed by cystatin C laboratory testing within 6 months of surgery

Exclusion Criteria:

* diagnosis of CKD stage 1 or 4-5
* home medications of angiotensin converting enzyme inhibitors (ACEi, such as lisinopril or captopril) or angiotensin receptor blocker (ARB, such as losartan, valsartan) diuretics, or trimethoprim
* IV contrast in last 30 days
* PMH of renal transplant, diabetes, hypertension, nephrotic syndrome or heart failure, asthma, or hyperthyroidism
* history of hyperkalemia
* recent glucocorticoid exposure
* procedure for oncologic indications
* ongoing viral or fungal infection, or chemotherapy
* allergy to NSAIDs

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of Acute Kidney Injury | From start of intervention, through 7 days later
  Acute kidney injury (AKI) will be assessed for according to Kidney Disease Improving Global Outcomes (KDIGO) criteria. Specifically, an AKI will be defined as a serum creatinine increase of ≥ 1.5 times baseline or ≥3 mg/dl increase, or a urine output <0.5ml/kg/h for 6 to 12 hours. While there are 3 stages of AKI, the investigators will consider AKI a binary outcome since all stages are managed the same clinically. Urine output is recorded as a routine part of strict intake & output monitoring by nursing. The serum creatinine will be compared to the pre-incisional/baseline data.

SECONDARY OUTCOMES:
Opiates received while inpatient | From start of intervention, through 7 days later
  Opiate use will be calculated as morphine equivalents per day, adjusted for weight.
Days with elevated pain score | From start of intervention, through 7 days later
  Pain scores will be assessed using the Faces Pain Scale - Revised (FPS-R) or the visual analogue scale (VAS) depending on age, per nursing routine. The former is used for patients aged 4-8 years, and latter for patients aged 9 and older. These have previously been shown to be interchangeable. Both pain scales have a range from 0-10, with 10 being the worst. This metric will not be captured for patients under 4 years of age. The percentage of days with severe, or a pain score greater than 7 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Rove, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ha D, Halstead NV, Blanchette ED, Wilcox DT, Vemulakonda VM, Wood DN, Rove KO. Risk of acute kidney injury after lower urinary tract reconstruction with early NSAID therapy: A propensity matched retrospective analysis. J Pediatr Urol. 2024 Oct;20(5):911-920. doi: 10.1016/j.jpurol.2024.07.005. Epub 2024 Jul 16. PMID 39089953